CLINICAL TRIAL: NCT00041730
Title: Phase II Trial of Rituxan(R) Plus FavId(TM) (Tumor-Specific Idiotype-KLH) and GM-CSF Immunotherapy in Patients With Grade 1 or 2 Follicular B-Cell Lymphoma
Brief Title: Rituxan Plus FavId (Idiotype Vaccine) for Low-grade Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Favrille (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FavId-04; NCT00060164 (obsolete NCT alias)
Record Dates: First submitted 2002-07-15; First posted 2002-07-17 (Estimated); Last update posted 2009-09-30 (Estimated); Status verified 2004-10

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: lymphoma; vaccine; idiotype; KLH; GM-CSF; FavId
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma

INTERVENTIONS:
Biological: Id-KLH

SUMMARY:
The purpose of this study is to evaluate the ability of patients treated with Rituxan® plus FavId™ and GM-CSF to mount an immune response (humoral and/or cellular) to KLH and their idiotype.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the ability of patients treated with Rituxan® plus FavId™ and GM-CSF to mount an immune response (humoral and/or cellular) to KLH and their idiotype. Secondary objectives are the determination of overall objective response rate, duration of response and time to progression. B-cell malignancies express a unique antigen, the immunoglobulin idiotype (Id), on their surface. Each B-cell harbors a unique genetic sequence used in production of unique Id protein. No normal B-cells possess that Id on their cell surface. Hence, Id protein should serve as an ideal target for individualized active immune therapy of NHL. Many of the antigens expressed by tumors (including Id) are only weak immunogens. To augment the immune response against Id, the Id protein must be chemically coupled to a strongly immunogenic protein. keyhole limpet hemocyanin (KLH) is a commonly used protein carrier capable of augmenting the body's immune reaction against Id protein. For vaccines which produce primarily an antibody response, there is a concern that combining immunotherapy with Rituxan®, which produces a rapid and sustained (up to 6 to 9 months post-treatment in 83% of patients) depletion of circulating and tissue-based B-cells, would blunt any antibody response. For vaccines that induce strong T-cell responses like Id-KLH plus GM-CSF, there is evidence in mice that depleting the host of B-cells could actually increase the T-cell response to the vaccine. GM-CSF is a hematopoietic growth factor that stimulates T-cell proliferation. T-cell response to both the patient's Idiotype and KLH will be measured during this trial.

ELIGIBILITY:
Inclusion Criteria

* 18 years of age or older
* Patients that are treatment naive OR
* Relapsed or refractory following chemotherapy OR
* Relapsed following a prior response to Rituxan(R) Note: Rituxan (R) may have been given as second-line therapy following an initial response to chemotherapy or in combination with chemotherapy for initial therapy of their disease.
* Tumor accessible for biopsy or previously existing recent biopsy material
* Measurable disease after node biopsy
* Histologically confirmed grade 1 or 2 follicular B-cell lymphoma (WHO classification)
* Performance status (ECOG) of 0, 1 or 2
* Absolute Granulocyte count > 1,000/mm3
* Platelets > 100,000/mm3
* Total Bilirubin <2 mg/dL
* AST and ALT <2x Upper Limit of Normal
* Creatinine < 1.5 mg/dL

Exclusion Criteria

* Patients who are refractory to Rituxan(R) Note: Patients who did not attain a CR or PR are considered to be refractory
* More than 2 prior treatment regimens (e.g. CHOP plus Rituxan(R) is one treatment regimen; CHOP followed by Rituxan(R) at initial relapse equals two treatment regimens)
* Treatment w/Fludarabine within 9 months of study entry
* Patients with > 5,000 lymphocytes
* Prior tumor-specific idiotype immunotherapy using the identical idiotype (patients whose idiotype has changed are eligible for retreatment with new idiotype)
* Concurrent immunosuppressive therapy (high-dose steroids; ect.)
* Known history of CNS lymphoma or meningeal lymphomatosis
* HIV positive
* Serious non-malignant disease (e.g., psychiatric disorders, compromised pulmonary function (e.g. active asthma, COPD, pneumonitis, bronchiolitis obliterans), congestive heart failure, or active uncontrolled bacterial, viral or fungal infections), or other conditions which, in the opinion of the investigator would compromise protocol objectives
* Prior malignancy (excluding non-melanoma carcinomas of the skin and in situ cervical carcinomas) unless in remission for >2 years
* Treatment with an investigational drug within 8 weeks prior to study entry
* Pregnant or nursing women NOTE: Women of childbearing potential should be advised to avoid becoming pregnant while receiving study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90
Dates: Start 2002-07

CONTACTS AND LOCATIONS:
Locations (15):
- United States (15):
  - University of California, San Diego, La Jolla, California
  - Tower Hematology Oncology Medical Group, Los Angeles, California
  - Oncology Associates of San Diego, San Diego, California
  - University California, San Francisco, San Francisco, California
  - University of Florida, Jacksonville, Jacksonville, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Chicago, Illinois
  - Ochsner Clinical Foundation, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - New York Medical College - Our Lady of Mercy Medical Center, Comprehensive Cancer Center, The Bronx, New York
  - Oncology/Hematology Care Clinical Cancer Institute, Cincinnati, Ohio
  - University Hospitals of Cleveland Case Western, Ireland Cancer Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - The Sarah Cannon Cancer Center, Nashville, Tennessee
  - University of Virginia, Charlottesville, Virginia